CLINICAL TRIAL: NCT03182569
Title: Use of a Flexible Catheter for the Administration of Subcutaneous Insulin in Diabetic Ketoacidosis
Brief Title: Flexible Catheter for Insulin in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGNPE-247-2016
Record Dates: First submitted 2017-03-14; First posted 2017-06-09 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetic Ketoacidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- flexible catheter (Experimental): The flexible Subcutaneous catheter for insulin administration
  Interventions: Device: FLEXIBLE CATHETER
- hourly rigid needle puncture (Active Comparator): Hourly rigid needle puncture for Subcutaneous insulin administration
  Interventions: Device: hourly rigid needle puncture

INTERVENTIONS:
Device: FLEXIBLE CATHETER
  Arms: flexible catheter
Device: hourly rigid needle puncture
  Arms: hourly rigid needle puncture

SUMMARY:
Use of a flexible subcutaneous catheter improves comfort in patients with DKA compared to the usual treatment with a metal needle.

DETAILED DESCRIPTION:
Assess whether the use of a flexible subcutaneous catheter improves comfort in patients with DKA compared to the usual treatment with a metal needle.

Compare the metabolic evolution of patients with DKA using a flexible subcutaneous catheter for insulin administration vs. a metal needle.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 5 to 18 years, admitted with diagnoses of DKA. DKA is defined when patients meets all the following biochemical baseline criteria (before initial hydration):
* Glucose> 200 mg / dl
* pH < 7.3
* Bicarbonate < 15mmol/l.

Exclusion Criteria:

* Patients referred from another institution with a different treatment, and those who requires intensive care on admission.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-11 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Comfort measured by a visual analogue scale for pain | between 10 to 14 hours
  Comfort measured by a visual analogue scale for pain (10cm = 0 meaning no pain and 10 meaning maximum pain) shown hourly after insulin administration until metabolic stability is achieved.

SECONDARY OUTCOMES:
Associated complications | 24 hours
  complications associated with the insulin administration device (local infection, extravasation)
Metabolic stability according to lab determinations | between 10 to 14 hours
  Time to reach the metabolic stability defined by: glycemia ≤250 mg/dl, pH ≥ 7.3, bicarbonate ≥ 15 mmol/L);

CONTACTS AND LOCATIONS:
Overall Officials: Laura Beaudoin, MD, Principal Investigator — Hospital General de Niños Pedro de Elizalde
Locations (1):
- Hospital General de Niños Pedro de Elizalde, Buenos Aires, Constitucion, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hanas R, Adolfsson P, Elfvin-Akesson K, Hammaren L, Ilvered R, Jansson I, Johansson C, Kroon M, Lindgren J, Lindh A, Ludvigsson J, Sigstrom L, Wiik A, Aman J. Indwelling catheters used from the onset of diabetes decrease injection pain and pre-injection anxiety. J Pediatr. 2002 Mar;140(3):315-20. doi: 10.1067/mpd.2002.122470. PMID 11953729
- [Derived] Beaudoin ML, Torrents M, Tittarelli MF, Hamui M, Ibarra M, Ferraro M, Ferreira JP. Use of a Flexible Catheter for the Administration of Subcutaneous Insulin in Diabetic Ketoacidosis: A Feasibility Controlled Clinical Trial. Hosp Pediatr. 2021 Apr;11(4):396-400. doi: 10.1542/hpeds.2020-0063. Epub 2021 Mar 9. PMID 33687988